CLINICAL TRIAL: NCT06213623
Title: Prevalence of an Early Success of Non-invasive Ventilation in the Emergency Departement. A Prospective Observational Study of the "Initiative Recherche Urgences" Network
Brief Title: Prevalence of an Early Success of Non-invasive Ventilation in the Emergency Departement.
Acronym: VENTIRU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VENTIRU
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Non Invasive Ventilation; Acute Respiratory Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-invasive ventilation is a mechanical ventilation who provides ventilatory support through a facemask, and without the need for tracheal intubation. In the emergency department, non-invasive ventilation is commonly used for the management of acute respiratory failure related with acute exacerbation of chronic obstructive pulmonary disease or with cardiogenic pulmonary oedema. Non-invasive ventilation is associated with an improvement in the outcomes, such as a decreasing in the intubation rate and in the mortality rate. Non-invasive ventilation failure is defined by a requirement to tracheal intubation in a patient managed by non-invasive ventilation. In the intensive care unit, non-invasive ventilation failure is reported from 15 to 50% of patients according to the ARF aetiologies. Due to delayed intubation, non-invasive ventilation failure is associated with poor outcomes and an increasing in the mortality rate. Due to the emergency department's patients (older and/or not to be intubate patients) the actual definition of non-invasive ventilation failure could not be applied as non-invasive ventilation may have been stopped not because it was unsuccessful but because it was unsuccessful in a patient with a do not intubate decision. Consequently, the prevalence of the absence of non-invasive ventilation success in the emergency department is unclear, and its predictive factor are unknown.

The aim is to measure the prevalence of the absence of non-invasive ventilation success in the emergency department. The secondary objective is to measure the association between an absence of non-invasive ventilation success and outcomes and to identify risk factor of an absence of non-invasive ventilation success in the emergency department.

It's a prospective observationnal multicenter study in department of Initiative Recherche Urgences Study Groups from January 2024, 15th to January 2024, 20th. The Initiative Recherche Urgences is a research network set up on the initiative of the Société Française de Médecine d'Urgence, with the aim of promoting and coordinating multicentre research projects in the field of emergency medicine, during short inclusion periods.

The primary outcome is the proportion of patients who do not have an early success of non-invasive ventilation. The investigators measure the absence of success instead of failure because failure is defined by intubation and most of patients managed with non-invasive ventilation in an emergency department will not be intubated because of their age. The absence of success is defined by at least one of the following criteria measured at 1-hour: death, cardiorespiratory arrest, tracheal intubation, respiratory rate over 30 breaths/min, neurological impairment defined by a Glasgow coma scale < 14, signs of increased work of breathing, haemodynamic failure (defined by mean arterial pressure < 65 mmHg despite volumetric expansion and/or catecholamines), early stop of non-invasive ventilation due to intolerance. The investigators choose to measure at one hour because non-invasive ventilation is provided from one to two hours in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or over 18 years old
* Patient admitted in an intrahospital or pre-hospital emergency department
* Patient managed with non invasive ventilation
* No objection to the use of data

Exclusion Criteria:

* Minors, incapacitated adults or patients deprived of their liberty.
* Patient with a care limitation, instruction not to be reanimated.
* Contraindication to initiation of nonninvasive ventilation at the start of management (non-COPD coma< 10 non-COPD, hemodynamic failure, incoercible vomiting)
* Patient who have low autonomy as defined by a WHO score ≥ 3 (bedridden for more than 50% of the day, not confined to it)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in an intrahospital or pre-hospital emergency department and managed with non invasive ventilation
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-01-27 (Estimated); Study Completion 2024-01-27 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who do not have an early success of non invasive ventilation | 1 hour
  The absence of success is defined by at least one of the following criteria measured at 1-hour: death, cardiorespiratory arrest, tracheal intubation, respiratory rate over 30 breaths/min, neurological impairment defined by a Glasgow coma scale < 14, signs of increased work of breathing, haemodynamic failure (defined by mean arterial pressure < 65 mmHg despite volumetric expansion and/or catecholamines), early stop of non invasive ventilation due to intolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie LESTIENNE, MD PHD, Principal Investigator — CHU Poitiers
Locations (1):
- Poitiers University Hospital, Poitiers, France

REFERENCES:
- [Derived] Marjanovic N, Lestienne J, Balen F, Coisy F, Gerlier C, Guenezan J, Mimoz O; SFMU-IRU network. Prevalence, risk factors and consequences of early clinical deterioration under non-invasive ventilation in emergency department patients: a prospective, multicentre, observational study of the French IRU Network. Crit Care. 2025 Jun 3;29(1):224. doi: 10.1186/s13054-025-05430-7. PMID 40462106